CLINICAL TRIAL: NCT03590184
Title: Cost-effectiveness Analysis Associated With the Use of Resorbable Biosynthetic Parietal Prostheses Compared to Biological Prostheses in Contaminated (mVHWG Grade 3) Abdominal Wall Reconstruction
Brief Title: Cost-effectiveness Analysis Between Biosynthetic and Biological Parietal Prostheses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7126
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Ventral Hernia
Keywords: Abdominal wall repair; Infection; Biologic mesh; Biosynthetic mesh; Cost-effectiveness
MeSH Terms: conditions — Hernia, Ventral; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with a biological prosthesis: patients who have received a biological prosthesis
- patients with a biosynthetic resorbable prosthesis: patients who have received a biosynthetic resorbable prosthesis

SUMMARY:
Eventration corresponds to the dehiscence of the abdominal wall, with passage of peritoneum and / or intra-abdominal viscera, through an acquired orifice of the abdominal wall. It is secondary to an old incision and occurs in 10 to 20% of cases after a laparotomy. At present, if there is no debate on the type of prosthesis to implant in case of clean surgery: it is a synthetic prosthesis. But in the case of contaminated surgery (modified Ventral Hernia Working Group grade 3), there is no consensus.

Since the 1990s, biological prostheses have been recommended, but they represent significant expenses for health facilities. They are very numerous, and their prices vary between 3 000 € and 12 000 €. The choice is therefore difficult for the surgeon.

In 2016 the Strasbourg University Hospital general surgery team made the choice to use biosynthetic prostheses. This attitude does not seem consensual and is not based on any recommendations at present, either in France or internationally. The homogenization of practices requires the availability of clinical and medico-economic data, particularly in view of the price differences that exist between different types of prostheses.

The main objective of this study will be to compare the use of biosynthetic prostheses with biological prostheses in the treatment of curative surgical treatment of mVHWG grade 3 incisional hernias in terms of cost and serious complications at 6 months.

The secondary objective of the study will be to estimate the number of early recurrences at 6 months avoided, thanks to the use of biosynthetic prostheses compared to biological prostheses.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* Patient who has consented to the use of her medical data for research purposes.
* emergency or planned surgery for an abdominal wall reconstruction, in the context of a contaminated surgery (mVHWG grade 3) at the CHU Strasbourg Hautepierre
* use of biological type (Cellis®, Xenmatrix®, Strattice®) or biosynthetic (Phasix®) parietal prostheses

Exclusion Criteria:

* Refusal of the patient to participate in the study
* prosthesis placed prophylactically, subcutaneously, endoscopically, for bridge

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - emergency or planned surgery for an abdominal wall reconstruction, in the context of a contaminated surgery (mVHWG grade 3) at the CHU Strasbourg Hautepierre
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness analysis | 6 months after surgery
  Cost-effectiveness Analysis Between Biosynthetic and Biological Parietal Prostheses

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Chirurgie générale et digestive, Strasbourg, France

REFERENCES:
- [Derived] Charleux-Muller D, Romain B, Boisson C, Velten M, Brigand C, Lejeune C. Cost-effectiveness analysis of resorbable biosynthetic mesh in contaminated ventral hernia repair. J Visc Surg. 2022 Aug;159(4):279-285. doi: 10.1016/j.jviscsurg.2021.06.001. Epub 2021 Jun 9. PMID 34116953